CLINICAL TRIAL: NCT05041244
Title: Identification of Biomarkers, Prognostic Indicators and Development of Novel Interface Devices for the Clinical Use of Topical Negative Pressure in Diabetic Wounds
Brief Title: Negative Pressure Wound Therapy in Diabetic Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mauritius (Other)
Collaborators: Ministry of Health and Wellness, Mauritius (Unknown); Higher Education Commission, Mauritius (Unknown); Acelity (Other)
Responsible Party: Principal Investigator, Archana BHAW LUXIMON, Professor, University of Mauritius
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 50/14.2.2018
Record Dates: First submitted 2021-08-30; First posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Diabetic Foot
Keywords: Negative pressure wound therapy, diabetic foot ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Superiority, multi-centre randomised parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional arm (Experimental): NPWT will be delivered through devices (ActiVac and InfoVac) according to FDA protocol in conjunction with the polyurethane foams. Dressing changed will be on a weekly basis.
  Interventions: Device: Negative pressure wound therapy delivered through VAC
- Control (Other): Standard of care Participants will be given the standard care provided in specialist foot care clinics or in-patients.
  Interventions: Device: Standard of care

INTERVENTIONS:
Device: Negative pressure wound therapy delivered through VAC — Initial cycle: Continuous first 48 hours Subsequent cycle: Consider intermittent DPC (5 min ON/2 mins OFF) for rest of the therapy Target Target Pressure: 50-175mmHg, to be titrated for more drainage Dressing change interval: every week; need for more frequent dressing need to be evaluated. More frequent change of adaptic can be considered. (Adaptic is a layer of thin dressing that will be in direct contact with the wound to reduce the risk of maceration and adherence to the dressing)
  Arms: Interventional arm
Device: Standard of care — Participants in the control arm will have their dressings changed as per the current standard of care.
  Effective management of DFU will depend on accurate diagnosis and assessment and appropriate debridement of non-viable tissues in patients from both arms Patients will be advised to continue off loading and any evidence of early infection should be promptly treated.
  Other Names: Hydrogel, foams, pad and other dressings
  Arms: Control

SUMMARY:
Topical Negative Pressure Wound Therapy (TNPW) is an established tool in the management of Diabetic foot ulcer in many countries. This treatment option is under utilized in the public sector of Mauritius. This study aims to determine the efficacy of TNPW through identification of biomarkers in the Mauritian setting compared with conventional treatment. Patient with DFU will be selected based on an eligible criteria and randomly assigned to intervention group or control group.

Primary Objective: To determine the efficacy of TNPW in the public sector in Mauritius Secondary Objectives: To compare healing times, prognostic factors skin biopsies based on biomarker, histological and genomic analysis A randomised controlled study is being proposed, where up to 100 participants will be recruited.

The wounds of participants in the intervention arm will be managed with 3 weeks of TNPW.

DETAILED DESCRIPTION:
Study Description: Topical Negative Pressure Wound Therapy (TNPW) is an established tool in the management of Diabetic foot ulcer in many countries. This treatment option is under utilized in the public sector of Mauritius. This study aims to determine the efficacy of TNPW through identification of biomarkers in the Mauritian setting compared with conventional treatment

Objectives:

Primary Objective: To determine the efficacy of TNPW in the public sector in Mauritius Secondary Objectives: To compare healing times, prognostic factors skin biopsies based on biomarker, histological and genomic analysis

Endpoints:

Primary Endpoint:

Incidence of complete wound closure at 7, 14 and 21 days Time for complete wound closure Side and depth of diabetic ulcer at 7, 14, 21 days Extent of granulation tissue (Epithelialisation) (7- 21 days)

Secondary Endpoints: Hospital stay, readmission, rate of amputation and rate of infections and adverse events Number of dressing changes

Study Population: 50 patients in each arm (interventional and control) Chronic diabetic ulcers, Wagner's 2-3 Male and female Diabetes Mellitus without renal and liver impairment Age 18- 74 years Stable patients with Diabetic foot ulcer A G Jeetoo Hospital, Port-Louis and Souillac District Hospital

Phase: 2 Description of Sites/Facilities Enrolling Participants: The study will take place at the above mentioned units Approval has been received by the Regional Health Director and Consultant in Charge and the Ministry of Health and Wellness for A G Jeetoo Hospital and Souillac District Hospital.

Patients will be recruited from the Diabetes Clinic or the General Surgery Department.

Patients with chronic diabetic ulcer fulfilling the eligibility criteria Description of Study Intervention: Patients will be randomized to Negative Pressure Wound Therapy (TNPW) arm and conventional treatment arm offered at the above named hospitals. TNPW devices will be used in patients in the intervention arm for 3 weeks.

TNPW is described as a medical procedure which involves application of a dressing to the wound. The dressing is attached to a vacuum device that provides sub-atmospheric pressures which help in the removal of exudates to promote the healing process. Dressings will be changed weekly.

Study Duration: 12 months Participant Duration: Each participant will be followed weekly during the procedure then 3 monthly to assess wound healing and enquire about need for further treatment including admissions and long term adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 - 75 years
4. In good general health as evidenced by medical history or diagnosed with diabetes mellitus or exhibiting signs of diabetic foot ulcers
5. Patients suffering from diabetic foot ulcer last more than 3 weeks
6. Patients with diabetes and presence of a foot wound for more than 3 weeks

Exclusion Criteria:

1. Patients under <18 years or above 75 years
2. Patients unable to provide consent
3. Patients suffering from chronic kidney disease or liver impairment or other chronic conditions
4. Patients on anticoagulants
5. Patients with non diabetic ulcers
6. Patients with severe peripheral vascular disease
7. Patients having contra-indication to negative pressure wound therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Wound closure | 3 weeks
  Any wound closure or % reduction in size

SECONDARY OUTCOMES:
Biomarkers | 3 weeks
  The amount of granulation will be determined macroscopically and microscopically through histology. Biomarkers such IL6 TNF and CD31/33 will be analysed from tissue specimens
complete wound closure | 1 year
  the incidence of complete closure will be determined and compared between the intervention group and the control group
Adverse events | 1 year
  Adverse events will include physical and psychological distress as well as infections and admissions to hospitals or recurrence of ulcer

CONTACTS AND LOCATIONS:
Overall Officials: Abha Jodheea-Jutton, MBBS MRCGP, Principal Investigator — University of Mauritius
Locations (1):
- University of Mauritius, Réduit, Moka District, Mauritius

IPD SHARING:
Plan to Share IPD: No
All IPD has been stored in digital format in anonymised way and might be shared with other researchers on request. The request will be considered by the members of the team.